CLINICAL TRIAL: NCT00789659
Title: Incisional Wound Vac in Obese Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI did not want to go forward with study at this time
Sponsor: University of Mississippi Medical Center (Other)
Collaborators: Orthopaedic Trauma Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2008-0142
Record Dates: First submitted 2008-11-12; First posted 2008-11-13 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2012-04

CONDITIONS: Wound Infection; Postoperative Complication
Keywords: Fracture fixation, internal; Obesity; Pelvis; Negative pressure wound therapy; Vacuum-assisted closure
MeSH Terms: conditions — Wound Infection; Postoperative Complications; Obesity | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VAC dressing (Experimental): The patients whose postoperative wound will be dressed with a negative pressure (V.A.C.) dressing.
  Interventions: Other: Negative pressure dressing

INTERVENTIONS:
Other: Negative pressure dressing — A completely occlusive dressing that is attached to a device that allows a constant negative pressure of 125 mmHg to be generated.
  Other Names: V.A.C.

SUMMARY:
It is the belief of the investigators that the current trends in complication rates associated with fixation of pelvic ring injuries and acetabular fractures in the obese are unacceptable. The overwhelming majority of these complications can be attributed to problems with surgical wound healing. The investigators feel that if a cost effective and easily performed intervention can be prospectively utilized in a specific at-risk orthopaedic trauma population in order to control a potentially devastating complication, then efforts in discovering such an intervention may prove valuable. It is our hypothesis that obese patients treated with V.A.C. therapy after standard closure of trauma-related, operative orthopaedic incisions will have fewer postoperative wound complications.

DETAILED DESCRIPTION:
Obesity has been shown to be an independent risk factor for postoperative surgical infections in a variety of obesity related and non-obesity related surgeries. With the risk of an increasingly more obese society, complication rates that significantly differ based on patients' relative obesity may become increasingly unacceptable. The purpose of the proposed prospective study is to evaluate the role that vacuum assisted closure (VAC) may play in reducing these complication rates. Negative pressure or vacuum assisted closure was first introduced in 1997 as a way to control and potentially treat chronic wounds. Since that time, the indications have exploded to include a variety of chronic and acute wound healing problems. We have anecdotally been using VAC therapy (V.A.C.;KCI, San Antonio, Texas) in an effort to control the postoperative draining that is nearly ubiquitous in our morbidly obese orthopaedic trauma patients. The V.A.C. dressing is applied to the acute postoperative wound and maintained during the immediate postoperative period. Although a novel approach to the use of the V.A.C., this use has been previously reported in the orthopaedic literature as a case series. To our knowledge, there has not been a prospective study evaluating the efficacy of the immediate placement of a V.A.C. dressing on postoperative wound infection rates in the setting of the morbidly obese orthopaedic trauma patient. It is our hypothesis that obese patients treated with V.A.C. therapy after standard closure of trauma-related, operative orthopaedic incisions will have fewer postoperative wound complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 - 64
* Patients with a BMI greater than or equal to 30
* Patients with acetabular, pelvic ring, or proximal femur fractures with a degree of displacement that would require an open reduction for treatment under normal circumstances

Exclusion Criteria:

* Patients not within variables defined by the inclusion criteria
* Abdominal or urological surgery during the same hospital admission
* Ipsilateral soft tissue injuries that can be classified as internal degloving injuries

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The comparative presence of drainage from the incisional wound treated with VAC therapy and the incisional wound treated with simple dry dressings at postoperative day 3. | 3 days

SECONDARY OUTCOMES:
The presence or absence of additional procedures needed to gain control of any wound complications. | 3 days
The amount of effluent contained in the V.A.C. canister. | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Graves, MD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

REFERENCES:
- [Background] Baugh N, Zuelzer H, Meador J, Blankenship J. Wound wise: wounds in surgical patients who are obese. Am J Nurs. 2007 Jun;107(6):40-50; quiz 51. doi: 10.1097/01.NAJ.0000271848.07721.24. PMID 17519604
- [Background] Canturk Z, Canturk NZ, Cetinarslan B, Utkan NZ, Tarkun I. Nosocomial infections and obesity in surgical patients. Obes Res. 2003 Jun;11(6):769-75. doi: 10.1038/oby.2003.107. PMID 12805398
- [Background] Falagas ME, Kompoti M. Obesity and infection. Lancet Infect Dis. 2006 Jul;6(7):438-46. doi: 10.1016/S1473-3099(06)70523-0. PMID 16790384
- [Background] Fleischmann E, Kurz A, Niedermayr M, Schebesta K, Kimberger O, Sessler DI, Kabon B, Prager G. Tissue oxygenation in obese and non-obese patients during laparoscopy. Obes Surg. 2005 Jun-Jul;15(6):813-9. doi: 10.1381/0960892054222867. PMID 15978153
- [Background] Karunakar MA, Shah SN, Jerabek S. Body mass index as a predictor of complications after operative treatment of acetabular fractures. J Bone Joint Surg Am. 2005 Jul;87(7):1498-502. doi: 10.2106/JBJS.D.02258. PMID 15995116
- [Background] Rubin RH. Surgical wound infection: epidemiology, pathogenesis, diagnosis and management. BMC Infect Dis. 2006 Nov 27;6:171. doi: 10.1186/1471-2334-6-171. PMID 17129369
- [Background] Wilson JA, Clark JJ. Obesity: impediment to postsurgical wound healing. Adv Skin Wound Care. 2004 Oct;17(8):426-35. doi: 10.1097/00129334-200410000-00013. PMID 15492679
- [Background] Argenta LC, Morykwas MJ, Marks MW, DeFranzo AJ, Molnar JA, David LR. Vacuum-assisted closure: state of clinic art. Plast Reconstr Surg. 2006 Jun;117(7 Suppl):127S-142S. doi: 10.1097/01.prs.0000222551.10793.51. PMID 16799380
- [Background] Morykwas MJ, Simpson J, Punger K, Argenta A, Kremers L, Argenta J. Vacuum-assisted closure: state of basic research and physiologic foundation. Plast Reconstr Surg. 2006 Jun;117(7 Suppl):121S-126S. doi: 10.1097/01.prs.0000225450.12593.12. PMID 16799379
- [Background] Venturi ML, Attinger CE, Mesbahi AN, Hess CL, Graw KS. Mechanisms and clinical applications of the vacuum-assisted closure (VAC) Device: a review. Am J Clin Dermatol. 2005;6(3):185-94. doi: 10.2165/00128071-200506030-00005. PMID 15943495
- [Background] Gomoll AH, Lin A, Harris MB. Incisional vacuum-assisted closure therapy. J Orthop Trauma. 2006 Nov-Dec;20(10):705-9. doi: 10.1097/01.bot.0000211159.98239.d2. PMID 17106382
- [Background] Porter SE, Russell GV, Dews RC, Qin Z, Woodall J Jr, Graves ML. Complications of acetabular fracture surgery in morbidly obese patients. J Orthop Trauma. 2008 Oct;22(9):589-94. doi: 10.1097/BOT.0b013e318188d6c3. PMID 18827587
- [Background] Porter SE, Graves ML, Qin Z, Russell GV. Operative experience of pelvic fractures in the obese. Obes Surg. 2008 Jun;18(6):702-8. doi: 10.1007/s11695-007-9320-y. Epub 2008 Mar 29. PMID 18373124